CLINICAL TRIAL: NCT06408675
Title: Loss of Cervical Lordosis an Association of Fibromyalgia Syndrome
Brief Title: Loss of Cervical Lordosis in Fibromyalgia Syndrome
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: B.10.1.TKH.4.34.H.GP.0.01/146
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Fibromyalgia, Cervical Lordosis
Keywords: Fibromyalgia, cervical lordosis
MeSH Terms: conditions — Fibromyalgia | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1 with a Cobb angle of ≤10°: cervical lordosis cobb angele ≤10°
  Interventions: Other: Visual Analog Scale (VAS), QOL (36-Item Short Form Survey (SF-36)), and Neck Disability Index (NDI) were used to assess pain, overall quality of life, functional disability respectively.
- group 2 with an angle greater than >10°: cervical lordosis cobb angele >10°
  Interventions: Other: Visual Analog Scale (VAS), QOL (36-Item Short Form Survey (SF-36)), and Neck Disability Index (NDI) were used to assess pain, overall quality of life, functional disability respectively.

INTERVENTIONS:
Other: Visual Analog Scale (VAS), QOL (36-Item Short Form Survey (SF-36)), and Neck Disability Index (NDI) were used to assess pain, overall quality of life, functional disability respectively. — Visual Analog Scale (VAS), QOL (36-Item Short Form Survey (SF-36)), and Neck Disability Index (NDI) were used to assess pain, overall quality of life, functional disability respectively.

SUMMARY:
Purpose: The causes of chronic and widespread pain in fibromyalgia (FMS) have not been eluciated yet. Previous reports determined that posture control changed, muscle strength decreased, body posture misaligned (maladaptive posture), and functional capacity decreased in FMS patients. The aim of this study was to investigate the relationship between loss of cervical lordosis, pain, quality of life (QOL) and neck disability in patients with FMS.

Methods: A total of 107 FMS (88 females and 20 males; range of age:18-65) were included to the study. Patients were divided into two groups according to the angle of cervical lordosis measured by the Cobb method, group 1 with a Cobb angle of ≤10°, and group 2 with an angle greater than >10°. Visual Analog Scale (VAS), QOL (36-Item Short Form Survey (SF-36)), and Neck Disability Index (NDI) were used to assess pain, overall quality of life, functional disability respectively.

ELIGIBILITY:
Inclusion Criteria:

Age range between 18 and 65

-Patients diagnosed with fibromyalgia according to the American College of Rheumatology 1990 criteria

Exclusion Criteria:

Patients diagnosed with known systemic (e.g., inflammatory rheumatic diseases, diabetes mellitus and systemic arterial hypertension), metabolic or endocrine diseasesas well as tumoral, neurologic or infectious diseases,

* Patients with a history of trauma and surgery affecting the neck area,
* Patients who received trigger point injection therapy for neck pain within the last 6 months,
* Patients with cervical disc herniation or myelopathy, spondylolisthesis, spondylolysis, cervicothoracic kyphoscoliosis,
* Patients who had been receiving therapy for any psychiatric diagnosis for the last 3 months and antidepressant drug use,
* Patients with history of neuropathic diseases,
* Patients with a condition affecting neck muscles, such as dystonia,
* Inflammatory muscle disease and myopathy
* Pregnant patients were not included to the study

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A total of 107 patients who applied to the physical therapy and rehabilitation outpatient clinic; . Age range between 18-65 , male-female, Patients diagnosed with fibromyalgia according to the American College of Rheumatology 1990 criteria
Sampling Method: Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | day 1,
  VAS scale used to measure the severity of pain (0-10 cm). According to this scale, the value 0 means no pain and the value 10 means very severe pain

SECONDARY OUTCOMES:
Quality of Life Scale-Short Form (SF-36) | day 1.
  This scale assesses many aspects of health and consists of 36 questions with 8 subtitles. The assessment is performed considering the last 4 weeks of the patient and the scale is assessed between 0 point and 100 points in which score 100 shows good health state, the score 0 shows poor health state
Neck disability index (NDI) | day 1
  This form has a total of 10 items, which includes pain severity, personal care, lifting, reading, headache, concentration, work status, driving, sleep and recreation. Scoring for each question ranges from 0 to 5 (0: the best health state and 5: the worst health state). High scores in patients mean serious disability. Total point were scored between 0 (no disability) and 100 (complete disability)

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara City Hospital, Ankara, Çankaya
  - Emine Esra Bilir, Ankara, Çankaya

IPD SHARING:
Plan to Share IPD: No